CLINICAL TRIAL: NCT06513169
Title: Lower Extremity Elevation to Minimize Hemodynamic Instability During Induction of General Anesthesia - a Prospective Randomized Controlled Study
Brief Title: Lower Extremity Elevation to Minimize Hemodynamic Instability During Induction of General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ranganathan Govindaraj, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-22-0145
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Post Induction Hypotension
Keywords: hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: LEE (Experimental)
  Interventions: Procedure: Group 1: LEE
- Group 2: no LEE (No Intervention)

INTERVENTIONS:
Procedure: Group 1: LEE — Patients will be in supine position during induction with a 12" wedge placed at the level of the Achilles tendon (LEE)
  Arms: Group 1: LEE

SUMMARY:
The purpose of this study is to determine if lower extremity elevation (LEE) will reduce the incidence of postinduction hypotension, to compare the utilization of vasoactive medications after induction in patients with LEE and patients without LEE and to determine if LEE will increase measured cardiac output

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA)3 or lower
* Patients requiring general anesthesia

Exclusion Criteria:

* Allergic reaction to drugs commonly used for general anesthesia including fentanyl, midazolam, propofol, ephedrine and phenylephrine
* Pregnant women
* Requiring rapid sequence induction
* Prisoners
* Patient refusal
* Emergency Surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants that demonstrate hypotension | From start of anesthesia upto institution of positive pressure ventilation (about 5 minutes)
  Hypotension is defined as the reduction in mean arterial pressure by 20% or greater comparing the blood pressure measured before induction of anesthesia

SECONDARY OUTCOMES:
Number of participants that demonstrate Nadir blood pressure | From start of anesthesia upto institution of positive pressure ventilation (about 5 minutes)
  Nadir blood pressure is the lowest value of blood pressure (BP) that can occur
Change in heart rate | From start of anesthesia upto institution of positive pressure ventilation (about 5 minutes)
Number of participants that need rescue vasoactive agents | From start of anesthesia upto institution of positive pressure ventilation (about 5 minutes)
Accumulated dose of rescue vasoactive agents | End of study (within 15 minutes of baseline)
Change in non-invasive cardiac output | From start of anesthesia upto institution of positive pressure ventilation (about 5 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Ranganathan Govindaraj, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No